CLINICAL TRIAL: NCT04444518
Title: The VAX-MOM Study: Increasing Influenza and Tdap Vaccination of Pregnant Women
Brief Title: Increasing Influenza and Tdap Vaccination of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Cynthia Rand, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005115
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Immunization; Infection; Pregnancy Related
Keywords: pertussis; influenza; vaccination; prenatal care
MeSH Terms: conditions — Infections; Whooping Cough; Influenza, Human | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAX-MOM Intervention (Experimental)
  Interventions: Behavioral: VAX-MOM Intervention
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: VAX-MOM Intervention — The multi-component VAX-MOM intervention will be comprised of: training in communication, provider prompts, standing orders, and feedback on vaccination rates.
  Arms: VAX-MOM Intervention
Behavioral: Standard of Care — Standard vaccine education and processes provided to patients by obstetric practices.
  Arms: Standard of Care

SUMMARY:
Pregnant women who get influenza are more likely than non-pregnant women to have serious complications, including hospitalizations, death, preterm labor and premature birth. Pertussis can cause hospitalization or death for newborns. However, influenza and Tdap vaccination rates for pregnant women are low nationally. In this study, the investigators will perform a randomized controlled trial aimed at practice change in obstetricians' offices, with an overall goal of reducing morbidity and mortality from influenza and pertussis infections.

DETAILED DESCRIPTION:
Infants under 6 months of age at increased risk of both influenza (flu) and pertussis disease, and pregnant women risk serious illness and premature labor from flu. The Advisory Committee on Immunization Practices recommends that women receive a flu vaccine in flu season, and tetanus toxoid, reduced diphtheria toxoid, acellular pertussis (Tdap) vaccine during each pregnancy (ideally between 27-36 weeks) to lower the risk for flu and pertussis disease for themselves and their infants. However, only half of pregnant women in the US receive a flu and Tdap vaccine, respectively; only 33% of women receive both vaccines. Lack of vaccination stems from a combination of patient (lack of knowledge, vaccine hesitancy), provider (suboptimal communication skills, missed opportunities), and system (e.g. lack of standing orders and patient reminders) factors. An effective intervention is needed to improve flu and Tdap vaccination rates for pregnant women. To address these low vaccination rates the investigators plan to use a clustered RCT (randomizing practices), allocating half of the participating practice sites within each health system to the VAX-MOM intervention and the other half to standard of care. The multi-component VAX-MOM intervention will be comprised of: training in communication, provider prompts, standing orders, and feedback on vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Sex is female
* Pregnant
* identified as being eligible for influenza or Tdap vaccine

Providers

* any provider, nurse or staff associated with the participating sites

Exclusion Criteria:

Patients

* none

Providers

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12760 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center (URMC), Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators upon request as part of a collaboration.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Practices
Period: Overall Study
Arm/Group | VAX-MOM Intervention | Standard of Care
Started | 5992; 12 Practices | 6768; 15 Practices
Completed | 5992; 12 Practices | 6768; 15 Practices
Not Completed | 0; 0 Practices | 0; 0 Practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAX-MOM Intervention | Standard of Care | Total
Number analyzed (Participants) | 5992 | 6768 | 12760
Age, Categorical [Count of Participants; unit: Participants] — Population: Regarding the counts for "Age, Categorical," date of birth (DOB) was unavailable in the EHR for 39 total subjects and thus, age could not be calculated. Due to this, 26 subjects have an unknown age in the "Intervention" group, and 13 subjects have an unknown age in the "Standard of Care" group.
  Participants
    number analyzed (Participants) | 5966 | 6755 | 12721
    <=18 years | 129 | 118 | 247
    Between 18 and 65 years | 5837 | 6637 | 12474
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5992 | 6768 | 12760
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 430 | 526 | 956
  Black | 694 | 1266 | 1960
  Hispanic | 547 | 721 | 1268
  White | 1831 | 2016 | 3847
  Unknown | 2490 | 2239 | 4729
Region of Enrollment [Number; unit: participants]
  United States | 5992 | 6768 | 12760

OUTCOME MEASURES:

1. Primary Outcome: Rate of Influenza Vaccination
Description: Influenza vaccination rate during pregnancy. Vaccination status will be obtained from patient electronic health records.
Time Frame: 10/1/2021-6/30/2022 (intervention flu season)
Population: Pregnant during flu season
Measure: Number; unit: participants
Arm/Group | VAX-MOM Intervention | Standard of Care
Number analyzed (Participants) | 4609 | 5294
participants | 2382 | 2496

2. Primary Outcome: Rate of Tdap Vaccination
Description: Tdap vaccination rate during pregnancy. Vaccination status will be obtained from patient electronic health records.
Time Frame: 7/1/2021 - 6/30/2022 (intervention period)
Population: Pregnant individuals during study period
Measure: Number; unit: participants
Arm/Group | VAX-MOM Intervention | Standard of Care
Number analyzed (Participants) | 5992 | 6768
participants | 4532 | 5452

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Arm/Group | VAX-MOM Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04444518/Prot_SAP_000.pdf